CLINICAL TRIAL: NCT04162457
Title: Effects of Caloric and Non-caloric Sweet Preloads on Neural Correlates of Physiological and Neurocognitive Responses in Healthy Participants
Brief Title: Mapping the 'Sweet Brain' in Healthy Participants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Manchester (Other)
Collaborators: Cargill (Industry)
Responsible Party: Principal Investigator, Nikoleta Stamataki, Chief Investigator, University of Manchester
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: 6814
Record Dates: First submitted 2019-11-11; First posted 2019-11-14 (Actual); Last update posted 2021-07-13 (Actual); Status verified 2021-07

CONDITIONS: Obesity; Sweeteners
MeSH Terms: conditions — Obesity | interventions — stevioside; Glucose; maltodextrin; Water

STUDY DESIGN:
Intervention Model Description: Counter-balanced, double-blind, crossover, within-subject design.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: This study is double blind. All participants are completing 4 testing sessions in randomised and counterbalanced order. Participants and researchers (who are also outcome assessors) are blinded to the beverages content. Un-blinding will be performed following analysis of results
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Stevia beverage (Experimental): Participants receive 4 study beverages in the 4 imaging sessions in randomised and counterbalanced order.
  Interventions: Dietary Supplement: Stevia
- Glucose beverage (Experimental): 330 ml of water with glucose (equal sweetness with the stevia beverage)
  Interventions: Dietary Supplement: Glucose
- Maltodextrin beverage (Experimental): 330 ml of water with maltodextrin (equal amount of calories as the glucose beverage)
  Interventions: Dietary Supplement: Maltodextrin
- Water (Placebo Comparator): 330 ml water
  Interventions: Dietary Supplement: Water

INTERVENTIONS:
Dietary Supplement: Stevia — Participants will be administered one of the study beverages at each one of the 4 imaging sessions.
  Arms: Stevia beverage
Dietary Supplement: Glucose — Participants will be administered one of the study beverages at each one of the 4 imaging sessions.
  Arms: Glucose beverage
Dietary Supplement: Maltodextrin — Participants will be administered one of the study beverages at each one of the 4 imaging sessions.
  Arms: Maltodextrin beverage
Dietary Supplement: Water — Participants will be administered one of the study beverages at each one of the 4 imaging sessions.
  Arms: Water

SUMMARY:
The human brain has a central role in regulating appetite and food intake. It integrates many metabolic, hedonic and trait-related signals that affect eating behaviour and determine when and how much we eat. The effects of non-nutritive sweeteners (NNS) that provide sweet taste with no calories on appetite, food intake thus weight status remain a subject of debate. In this study, the investigators aim to investigate whole brain response to the ingestion of beverages sweetened with caloric sugars (glucose, maltodextrin) or NNS (stevia) as well as neural substrates of attentional bias to food (pre-and post consumption) in healthy lean participants.

DETAILED DESCRIPTION:
Non-nutritive sweeteners (NNS) are zero or no calorie alternatives to caloric sugars and their role in appetite and weight status remains inconclusive. NNS similarly as caloric sweeteners activate the oral sweetness receptors and conscious perception of sweetness. However caloric sugars and NNS differ in their metabolic fate after ingestion, so that caloric sugars lead to raised blood glucose, insulin and satiety inducing gut-peptide levels after meals, but NNS do not influence postprandial metabolism. A recently proposed model suggests that metabolic signals may have indirect effects on food reward processing via alterations in higher cognitive function such as attention (Higgs et al. 2017), the role of sweetness in this model is yet to be examined.

In the proposed study stevia-sweetened beverage will be used as the NNS, glucose-sweetened beverage as the caloric sweetener, water as a non-sweet non-caloric control and maltodextrin as a non-sweet caloric control. The study has two aims: first to investigate whole brain responses following the oral consumption of caloric sugars versus NNS using and physiological MRI, and second to examine the neural correlates of the attentional bias to food cues following the consumption of caloric sugars- vs. NNS-sweetened beverages using task-based functional Magnetic Resonance Imaging (fMRI).

In this study participants will be asked to come to the imaging facility on four separate occasions, corresponding to the four study beverages, glucose, stevia, maltodextrin and water. Before coming to an imaging session participants should consume a breakfast of their preference at home (which will be repeated before each session) and then fast for 3-4 hours. Upon arrival subjects will fill in their mood ratings, and the breakfast composition questionnaire and will be ready to start. Firstly, neural responses will be measured (before consumption of the study beverages) while subjects perform a food visual dot probe task (VPT) previously validated to show differences in attentional bias to food between fasted and fed states (Stamataki et al. 2019). Secondly, a physiological MRI measurement will be performed (Little et al. 2013) which will last 40 minutes. Third, subjects will perform again the VPT (after the consumption of the study beverage) whilst an fMRI measurement will be performed.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 - 40 years
* BMI between 18.5-25 kg/m2
* Registered to a GP
* Non-restrained eaters, restraint eating score on the Dutch Eating Behaviour Questionnaire (DEBQ) ≤ 3
* Healthy - general good health
* Currently not taking any medication (other than females taking the oral contraceptives or over the counter medication such as paracetamol)
* Normal or corrected vision
* Right-handedness (including left-handers could bias the results because of the laterality of brain functions)
* Regular breakfast eaters (≥5 times per week)
* Stable weight, ± 5 kg last 3 months
* No self-reported food allergy or intolerance to foods supplied during the study
* No or low NNS consumers (up to 1 can of diet soda per week or 1 sachet of NNS per week)
* Willing to comply with the study protocol
* Willingness to be informed about chance findings of pathology
* The participant is capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form.
* The participant is able to read, comprehend and record information written in English.
* A signed and dated written informed consent is obtained from the participant.

Exclusion Criteria:

* Habitual NNS consumers, >1 can of diet beverage or >1 table packet of sweeteners per week
* Subjects who have a non-removable metal object in or at their body, such as, for example: heart pace-maker, artificial heart valve, metal prosthesis, implants or splinters, non-removable dental braces
* Tattoos, that are older than 15 years
* Claustrophobia
* Pathological hearing ability or an increased sensitivity to loud noises
* Operation less than 3 months ago
* Acute illness or infection during the last 4 weeks
* Moderate or severe head injury
* Any metabolic (e.g. metabolic disorder, diabetes, insulin resistance), psychological (e.g. depression), gastrointestinal or neurological (e.g. epilepsy, headache disorder, multiple sclerosis, traumatic brain injuries) diseases or medication in relation to these diseases.
* Currently experiencing anxiety or depression
* Use of recreational substances in the last month
* Age under 18 years or over 40 years old.
* BMI >25 kg/m2 and <18.5 kg/m2
* Restrained eaters (DEBQ for restraint eating ≥ 3)
* Current weight loss regimens, or more than 5 kg weight loss/gain in the last 3 months
* Subjects who follow special diets for weight maintenance, such as Atkins Diet, Weight Watchers, gluten-free diet, The Zone diet, Vegetarian Diet, Raw Food Diet etc.
* Subjects having breakfast less than 5 times per week.
* Eating disorders (binge eating disorder, bulimia etc)
* Current or past history of drug or alcohol dependency - alcohol consumption exceeding 14 units a week
* Female participants who are, or may be, pregnant, or currently lactating.
* Subjects who regularly consume dietary supplements for weight loss, muscle building etc.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2019-11-14 (Actual); Primary Completion 2021-03-31 (Actual); Study Completion 2021-03-31 (Actual)

PRIMARY OUTCOMES:
physMRI whole brain responses to stevia, glucose and maltodextrin | -10 minutes to 30 minutes post consumption
  Participants will undergo a physiological MRI, which will include 10 minutes of baseline (resting), 10 minutes of drinking the solution, and 20 minutes post-consumption (resting).
fMRI brain response while performing a food visual dot probe task (VPT) | 10 minutes (twice)
  Before and 30 minutes after the consumption of the study beverage, participants will perform a food VPT which is designed to assess attentional bias to food cues while an fMRI will be conducted.
  Subjects neural activation when they are responding to congruent trials (dot appearing on the position of a food picture) compared to incongruent trials (dot appearing on the position of a neutral picture).

SECONDARY OUTCOMES:
Attentional bias to food cues (behavioral) | pre- and post (30 minutes) consumption of the study beverage
  Reaction times to congruent and incongruent trials will be recorded, and an attentional bias to food cues score will be calculated and expressed as the difference pre-and post consumption across the 4 experimental conditions.
Appetite ratings | -10 minutes (before consumption) to 30 minutes post-consumption
  Participant will be asked to rate their subjective appetite (hunger, fullness) at regular intervals during the physMRI. The mean ratings over time, change from baseline as well as area under the curve will be assessed.
  Scale includes 0-10 values where 0 is not at all (i.e. not hungry at all) and 10 is extremely (i.e. extremely hungry)
Sweetness ratings | at 10 minutes postprandially
  Following the consumption of the beverages participants will be asked to rate the sweetness of the beverage they consumed.
  Scale includes 0-10 values where 0 is not at all (i.e. not sweet at all) and 10 is extremely (i.e. extremely sweet)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Manchester, Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual Participant Data (IPD) will be shared in an open data repository, provided participants consent.
Time Frame: Data will become available after the results of the study will get accepted for publication by an international peer-reviewed journal, provided participants consent.
Access Criteria: All researchers

REFERENCES:
- [Background] Stamataki NS, Elliott R, McKie S, McLaughlin JT. Attentional bias to food varies as a function of metabolic state independent of weight status. Appetite. 2019 Dec 1;143:104388. doi: 10.1016/j.appet.2019.104388. Epub 2019 Jul 31. PMID 31376438
- [Background] Little TJ, McKie S, Jones RB, D'Amato M, Smith C, Kiss O, Thompson DG, McLaughlin JT. Mapping glucose-mediated gut-to-brain signalling pathways in humans. Neuroimage. 2014 Aug 1;96:1-11. doi: 10.1016/j.neuroimage.2014.03.059. Epub 2014 Mar 28. PMID 24685436